CLINICAL TRIAL: NCT03718624
Title: A Study of Intraperitoneal and Intravenous Paclitaxel Plus Apatinib and S-1 Conversion Therapy for Gastric Cancer With Positive Exfoliative Cancer Cells
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hebei Medical University (Other)
Responsible Party: Principal Investigator, Qun Zhao, Principal Investigator, Hebei Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HRA-G03
Record Dates: First submitted 2018-10-23; First posted 2018-10-24 (Actual); Last update posted 2018-10-31 (Actual); Status verified 2018-10

CONDITIONS: Gastric Cancer With Positive Exfoliative Cancer Cells
MeSH Terms: interventions — apatinib; Paclitaxel; S 1 (combination)

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- paclitaxel,apatinib and S-1 (Experimental)
  Interventions: Drug: apatinib; Drug: paclitaxel; Drug: S-1

INTERVENTIONS:
Drug: apatinib — apatinib：500mg qd po, 28 days is a cycle. preoperative 2 cycles, 2 cycles after surgery.
Drug: paclitaxel — Paclitaxel: intraperitoneal paclitaxel 20 mg/m2 and intravenous paclitaxel 50 mg/m2 on days 1 and 8 ，21 days is a cycle. preoperative 3 cycles, 3 cycles after surgery.
Drug: S-1 — S-1： According to the body surface area, BSA <1.25m2，40mg bid; 1.25m2≤BSA≤1.5m2，50mg bid; BSA >1.5m2, 60mg bid. Take the medicine twice daily for 2 weeks, then suspend for 1 week. preoperative 3 cycles, 3 cycles after surgery.

SUMMARY:
The purpose of this study is to investigate the efficacy and safety of intraperitoneal and intravenous paclitaxel plus apatinib and S-1 in the conversion therapy of gastric cancer with positive exfoliative cancer cells

ELIGIBILITY:
Inclusion Criteria:

1. Untreated (e.g. chemotherapy, radiotherapy and other antitumor therapy);
2. Age:18 to 70 years old;
3. Man or female (except pregnant and lactating women);
4. Confirmed to gastric adenocarcinoma;
5. Proven gastric cancer of T stage was T3 and T4, and no distant metastasis was observed. The exfoliative cancer cells detection in peritoneal washes was positive;
6. Blood cell count has to meet the following criteria:

   WBC≥3.5×109/L; ANC≥1.5×109/L; PLT≥100×109/L; HB≥90g/L;
7. Liver/kidney function has to meet the following criteria:

   ALT and AST≤2.5*ULN TBIL<1.5*ULN； Serum creatinine ≤1.5*ULN;
8. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1;
9. Participants were willing to join in this study, good adherence and written informed consent.

Exclusion Criteria:

1. Patients with other malignant tumors within 5 years;
2. Metastasis was found to be visible to the naked eye;
3. It has serious or uncontrolled heart diseases and infections (Including atrial fibrillation, angina pectoris, cardiac insufficiency, ejection fraction less than 50%, poor-controlled hypertension and so on);
4. History of psychiatric drugs abuse and can't quit or patients with mental disorders;
5. Patients with severe or uncontrollable mental illness;
6. Patients with tendency of gastrointestinal bleeding, including the following: a local active ulcerative lesions, and defecate occult blood (+ +).Has melena and hematemesis in two months;
7. Pregnant or lactating women;
8. It have serious harm to the patient's safety or affect the patients who have completed the research.
9. The researchers think inappropriate.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2018-10-30 (Estimated); Primary Completion 2019-10-30 (Estimated); Study Completion 2020-10-30 (Estimated)

PRIMARY OUTCOMES:
R0-resection rate | within 3 weeks after surgery
  There was no residual by the microscope
Conversion to negative rate | within 3 weeks after surgery
  Exfoliative cytology positive gastric cancer conversion to negative rate.

SECONDARY OUTCOMES:
Overall survival (OS) | 5years
  Baseline to measured date of death from any cause
Progression free survival (PFS) | 5years
  Baseline to measured date of progression or death from any cause
Adverse events | 5 years
  Toxicity according to the Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0.The number of Participants with adverse events will be recorded at each treatment visit.